CLINICAL TRIAL: NCT04992585
Title: Primary Versus Secondary Metal Stent Implantation in PTBD in Patients With Extrahepatic Malignant Bile Duct Obstruction
Brief Title: Primary Versus Secondary Metal Stent Implantation in PTBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theresienkrankenhaus und St. Hedwig-Klinik GmbH (Other)
Collaborators: Universitätsmedizin Mannheim (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PTBD retro 002
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2021-08-12 (Actual); Status verified 2021-08

CONDITIONS: Bile Duct Obstruction; Extrahepatic Cholestasis
Keywords: Bile Duct Obstruction; Self Expandable Metallic Stents
MeSH Terms: conditions — Cholestasis; Cholestasis, Extrahepatic

STUDY DESIGN:
Intervention Model Description: Retrospective comparison of two similar interventions with small modification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PTBD with primary metal stent implantation (Experimental): PTBD with primary metal stent implantation is performed in the same session as a one step-procedure
  Interventions: Device: Percutaneous transhepatic implantation of self-expandable metal stent
- PTBD with secondary metal stent implantation (Active Comparator): PTBD with secondary metal stent implantation is performed as a two step-procedure with metal stent implantation 3 to 7 days after previous percutaneous transhepatic biliary drainage and insertion of a plastic catheter
  Interventions: Device: Percutaneous transhepatic implantation of self-expandable metal stent

INTERVENTIONS:
Device: Percutaneous transhepatic implantation of self-expandable metal stent — A self-expandable metal stent is inserted into the extrahepatic bile duct which is obstructed by malignant disease

SUMMARY:
The aim is to compare percutaneous transhepatic biliary drainage (PTBD) with primary metal stent implantation (one stage-procedure) with PTBD with secondary metal stent implantation in terms of adverse events.

DETAILED DESCRIPTION:
Percutaneous transhepatic biliary interventions (PBI) are used in biliary tract diseases when endoscopic access was not successful or not possible due to anatomical changes after abdominal surgery. Self-expandible metal stents (SEMS) can be applied percutaneously in patients with malignant extrahepatic bile duct obstruction. In this setting, PTBD is usually performed as a two step-procedure with primary drainage of the accumulated bile fluid by an external or an external/internal plastic stent and a secondary metal stent implantation at an interval of a few days. PTBD with primary metal stent implantation might shorten the hospital stay and is therefore equal to the increasingly used method of endoscopic ultrasound-guided biliary drainage (EUS-BD). EUS-BD offers a one step-procedure with primary metal stent implantation which is probably associated with lesser adverse events (AE) than PTBD with secondary metal stent implantation. However, it is not clear whether PTBD with primary metal stent implantation shows fewer adverse events than PTBD with secondary stent implantation. The aim of this study is to retrospectively analyze the prospectively collected data of PTBDs with primary or secondary metal stent implantation in patients with proximal and distal malignant bile duct obstruction. The focus of this single center study will be to compare the two approaches in terms of adverse events. Adverse events in PTBD might range from very mild to fatal. Therefore, the severity of the adverse events has been considered in the calculation.

ELIGIBILITY:
Inclusion Criteria:

* PTBD with metal stent implantation into the extrahepatic bile duct
* malignant and non-resectable extrahepatic bile duct obstruction

Exclusion Criteria:

* benign extrahepatic bile duct obstruction

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Adverse events | From the intervention until 30 days after
  All adverse events which have been documented in the medical record were analyzed and classified as mild, moderate, severe or fatal/death according to the AE severity grading system of the American Society of Gastrointestinal Endoscopy (ASGE)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Schmitz, MD, Principal Investigator — Theresienkrankenhaus Mannheim, University of Heidelberg
Locations (1):
- Tertiary referral hospital: Theresienkrankenhaus und St. Hedwig Hospital, Academic, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharaiha RZ, Khan MA, Kamal F, Tyberg A, Tombazzi CR, Ali B, Tombazzi C, Kahaleh M. Efficacy and safety of EUS-guided biliary drainage in comparison with percutaneous biliary drainage when ERCP fails: a systematic review and meta-analysis. Gastrointest Endosc. 2017 May;85(5):904-914. doi: 10.1016/j.gie.2016.12.023. Epub 2017 Jan 4. PMID 28063840
- [Background] Venkatanarasimha N, Damodharan K, Gogna A, Leong S, Too CW, Patel A, Tay KH, Tan BS, Lo R, Irani F. Diagnosis and Management of Complications from Percutaneous Biliary Tract Interventions. Radiographics. 2017 Mar-Apr;37(2):665-680. doi: 10.1148/rg.2017160159. PMID 28287940
- [Background] Cotton PB, Eisen GM, Aabakken L, Baron TH, Hutter MM, Jacobson BC, Mergener K, Nemcek A Jr, Petersen BT, Petrini JL, Pike IM, Rabeneck L, Romagnuolo J, Vargo JJ. A lexicon for endoscopic adverse events: report of an ASGE workshop. Gastrointest Endosc. 2010 Mar;71(3):446-54. doi: 10.1016/j.gie.2009.10.027. No abstract available. PMID 20189503